CLINICAL TRIAL: NCT06350305
Title: Screening Study at High-risk Chronic Obstructive Pulmonary Disease
Brief Title: Screening for High-risk Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Screening for high-risk COPD
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: High-risk COPD
Keywords: high-risk COPD; scale
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire survey — subjects fill out questionnaires

SUMMARY:
This study is a multicenter cross-sectional study design aimed at screening risk factors for the combination of disease and syndrome in high-risk individuals with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Targeting high-risk populations for chronic obstructive pulmonary disease (COPD), targeted at key issues such as unclear risk factors and lack of prevention and treatment plans, high-risk population screening was conducted to identify risk factors. This study is expected to detect at least 3600 high-risk individuals with early-stage chronic obstructive pulmonary disease. The incidence rate of high-risk individuals in the early stage of chronic obstructive pulmonary disease is 30%, which means the total screening population is 12000 cases.

ELIGIBILITY:
Inclusion Criteria:

* According to the Diagnosis and Treatment Guidelines for Chronic Obstructive Pulmonary Disease (Revised in 2021), a multi-stage cluster random sampling method was used to select individuals from representative administrative villages with a history of chronic cough or sputum production, breathing difficulties, recurrent lower respiratory tract infections, and/or exposure to potential risk factors for chronic obstructive pulmonary disease.
* The investigators agreed to participate in this clinical study by voluntarily signing an informed consent form.

Exclusion Criteria:

* Patients who are delirious, have impaired consciousness, dementia, various psychiatric disorders, etc., and cannot be accurately informed of their basic physical condition.
* Patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the Diagnosis and Treatment Guidelines for Chronic Obstructive Pulmonary Disease (Revised in 2021), a multi-stage cluster random sampling method was used to select individuals from representative administrative villages with a history of chronic cough or sputum production, breathing difficulties, recurrent lower respiratory tract infections, and/or exposure to potential risk factors for chronic obstructive pulmonary disease.
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
COPD screening questionnaire from Terrassa (EGARPOC) | During screening
  3-29 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥13, the participant needed to be seen by a physician for further testing to determine if they had COPD.
COPD assessment in primary care to identify undiagnosed respiratory disease and exacerbation risk questionnaire (CAPTURE) | During screening
  0-6 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥2, the participant needed to be seen by a physician for further testing to determine if they had COPD.
COPD Assessment Test (CAT) | During screening
  0-40 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was >10, the participant needed to be seen by a physician for further testing to determine if they had COPD.
COPD screening questionnaire (COPD-Q) | During screening
  0-10 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥4, the participant needed to be seen by a physician for further testing to determine if they had COPD.
chronic obstructive pulmonary disease diagnostic questionnaire (CDQ) | During screening
  0-38 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥17, the participant needed to be seen by a physician for further testing to determine if they had COPD.
modified chronic obstructive pulmonary disease diagnostic questionnaire (mCDQ) | During screening
  0-45 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥18, the participant needed to be seen by a physician for further testing to determine if they had COPD.
Simple screening questionnaire | During screening
  0-11 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥6, the participant needed to be seen by a physician for further testing to determine if they had COPD.
lung function questionnaire (LFQ) | During screening
  5-25 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≤18, the participant needed to be seen by a physician for further testing to determine if they had COPD.
chronic obstructive pulmonary disease screening questionnaire (COPD-SQ) | During screening
  0-38 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥16, the participant needed to be seen by a physician for further testing to determine if they had COPD.
chronic obstructive pulmonary disease population screener questionnaire (COPD-PS) | During screening
  0-10 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥5, the participant needed to be seen by a physician for further testing to determine if they had COPD.
Chronic Obstructive Pulmonary Disease Risk Scale (COPDRS) | During screening
  0-9 scores. Scores for each questionnaire item were tallied based on the participant's responses, and if the total score was ≥5, the participant needed to be seen by a physician for further testing to determine if they had COPD.
Standardised Scale of Physical Fitness in Chinese Medicine | During screening
  Answer all the questions in the Classification and Determination of Physical Qualities in Chinese Medicine Table. Each question is rated on a 5-point scale, and the raw and transformed scores are calculated to determine the type of physical qualities according to the criteria. Raw score = sum of the scores of each entry. Transformation score = [(raw score - number of entries)/(number of entries × 4)] × 100.
Syndrome therapeutic evaluation scale of chronic obstructive pulmonary disease (COPD-STES) | During screening
  Subjects should fill in the relevant entries truthfully according to the category of symptoms as judged by the doctor and tick the appropriate box. Among them, the part of tongue and pulse should be filled in by the doctor.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China